CLINICAL TRIAL: NCT05037981
Title: Evaluation of Early Systemic Stabilization Therapy on Recent Onset Localized Non-segmental Vitiligo
Brief Title: Effect of Early Systemic Stabilization Therapy on Recent Onset Vitiligo
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Saadi, Dr, Cairo University
Other Study IDs: vit105
Record Dates: First submitted 2021-09-03; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vitiligo is a distressing disorder of depigmentation. In spite of multiple successful therapeutic regimens, disease relapse remains a challenge to patients and physicians. Most guidelines consider systemic treatments only in rapidly progressive disease with wider surface areas. This delay in halting the immune attack, may give the chance for further disease progression as well as establishment of resident memory T cell population predisposing to future disease relapses. The aim of this study was to assess the ability of early systemic therapy of localized (<2% BSA), recent onset (<6 months) vitiligo to control disease activity and minimize the possibility of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 6 years old of both genders
* Early onset vitiligo (˂6m duration)
* Body surface area (BSA) affected ≤2%

Exclusion Criteria:

* Patients who received any previous treatment for vitiligo
* Pregnant and lactating females
* Patients with other cutaneous or systemic autoimmune diseases
* Patients with contraindication to systemic corticosteroids

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with active localized vitiligo
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-10-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Duration needed to arrest of vitiligo activity | 6 months
  Time needed for vitiligo patients to stop developing new lesions of vitiligo
Duration of maintaining vitiligo stability | 5 years
  Time before any new vitiligo lesions reappear

CONTACTS AND LOCATIONS:
Overall Officials: Samia Esmat, MD, Principal Investigator — Cairo University; Rania Mogawer, MD, Principal Investigator — Cairo University; Dalia Bassiony, MD, Study Director — Cairo University; Suzan Shalaby, MD, Study Chair — Cairo University; Rehab Hegazy, MD, Study Chair — Cairo University; Nanis Ragab, MD, Study Chair — Cairo University; Sarah Ibrahim, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No
Sharing in published manuscript in a journal